CLINICAL TRIAL: NCT01677260
Title: A Combined Single Dose Study Under Fasting Condition And Multiple Doses Study Under Normal Diabetic Meal Comparing the Bioavailability of Two Formulations of 500 mg Metformin Hydrochloride Extended Release Tablets.
Brief Title: Bioequivalence Study of Two Formulations of 500 mg Metformin Extended Release Tablet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PR. 143/EQL/2009
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Metformin XR BE Study in Healthy Volunteers With Single and Multiple Dose
Keywords: Biguanide; anti-hyperglycaemic; bioavailability; bioequivalence; metformin; pharmacokinetics
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): 500 mg metformin hydrochloride extended release caplet (PT Ferron Par Pharmaceuticals)
  Interventions: Drug: 500 mg metformin hydrochloride extended release caplet (test drug)
- Group II (Active Comparator): 500 mg metformin hydrochloride prolonged release tablet (PT Merck Pharmaceuticals)
  Interventions: Drug: 500 mg metformin hydrochloride prolonged release tablet (reference drug)

INTERVENTIONS:
Drug: 500 mg metformin hydrochloride extended release caplet (test drug) — In each of the two study periods (separated by a washout of one week) a single and multiple dose of test or reference product was administered.
  Other Names: Glumin® XR, manufactured by PT Ferron Par Pharmaceuticals
  Arms: Group I
Drug: 500 mg metformin hydrochloride prolonged release tablet (reference drug) — In each of the two study periods (separated by a washout of one week) a single and multiple dose of test or reference product was administered.
  Other Names: Glucophage® SR, manufactured by PT Merck Pharmaceuticals
  Arms: Group II

SUMMARY:
This was a single centre, single-blind, randomized, balanced, combined single dose study under fasting condition and multiple doses study under fed condition with normal diabetic-meal, two-period, two-sequence cross-over study to to compare the bioavailability of metformin hydrochloride 500 mg extended release caplet (test drug) and metformin hydrochloride 500 mg prolonged release tablet (reference formulation).

DETAILED DESCRIPTION:
On Day 1, to obtain pharmacokinetic profile of a single dose, the test or reference drugs were given with 200 mL of water and swallowed without chewing the drug. For multiple doses administration at Day 2 until Day 5, the study drugs were administered at a regimen of one tablet each day, 30 minutes after breakfast. Time of drug administration was standardized for all participating subjects throughout the study period.

From each subject, on Day 1 until Day 5 blood samples were drawn 5 mL before breakfast and drug administration; and breakfast was provided only on Day 2 until Day 5. Only on Day 1 and Day 5 after drug administration, the blood samples were drawn 5 mL each at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 10, 12, 16 and 24 hours.

The blood samples drawn on Day 1 were used to show the single dose pharmacokinetic profile under fasting condition; while those drawn on Day 5 were used to show the multiple-dose-pharmacokinetic profile after meal intake.

One week after the first drug administration (washout period), the same procedure was repeated with the alternate drug.

The plasma concentrations of metformin were determined by high performance liquid chromatography with ultraviolet detection (HPLC-UV). The pharmacokinetic parameters assessed in the single dose study were AUCt, AUCinf, Cmax, tmax, and t1/2. The pharmacokinetic parameters assessed in multiple doses study at steady state phase were AUCtau, Cmax, Cmin, and t1/2.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with absence of significant diseases or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening.
* Age of 18 - 55 years
* Preferably non-smokers or smoke less than 10 cigarettes per day
* Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study.
* BMI 18 - 25 kg/m2
* Vital signs (after 10 minutes rest) were within the following ranges:
* SBP 100 - 120 mmHg
* DBP 60 - 80 mmHg
* Pulse rate 60 - 90 bpm

Exclusion Criteria:

* Personal/family history of allergy or hypersensitivity or contraindication to metformin hydrochloride or other biguanides and allied drug.
* Pregnant or lactating women and women of childbearing potential without adequate contraception
* Any major illnesses in the past 90 days or clinically significant ongoing chronic medical illnesses
* Clinically significant illness within 4 weeks prior to the administration of study medication
* Presence of any clinically significant abnormal values during screening
* Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV
* Clinically significant haematology abnormalities
* Clinically significant electrocardiogram (ECG) abnormalities
* Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug
* History of drug (cocaine, amphetamines, opiates, cannabis) or alcohol abuse within 12 months prior to screening for this study
* Participation in any clinical trial within the past 90 days
* History of any bleeding or coagulative disorders
* History or presence of asthma bronchial or related bronchospastic conditions
* History of seizures, epilepsy or any kind of neurological disorders
* History of difficulty with donating blood or difficulty in vein puncture of left or right arm
* A donation or loss of 500 mL (or more) of blood within 3 months before this study's first dosing day
* Intake of any prescription or non-prescription drugs, food supplements or herbal medicines within 14 days of this study's first dosing day
* Any food allergy, intolerance, restriction or special diet that in the opinion of the Research Physician, could contraindicate the subject's participation in this study
* Any reason in the opinion of the Research Physician, would prevent the subject from participating in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 24 hours
  Relative bioavailability (primarily measured by AUC and Cmax) between metformin hydrochloride 500 mg extended release caplet (test formulation) and metformin hydrochloride 500 mg prolonged release tablet (reference formulation) at a single dose.
Bioavailability | 5 days
  Relative bioavailability (primarily measured by AUC and Cmax) between metformin hydrochloride 500 mg extended release caplet (test formulation) and metformin hydrochloride 500 mg prolonged release tablet (reference formulation)at multiple doses.

SECONDARY OUTCOMES:
Bioavailability | 24 hours
  Relative bioavailability (secondarily measured by tmax and t1/2) between metformin hydrochloride 500 mg extended release caplet (test formulation) and metformin hydrochloride 500 mg prolonged release tablet (reference formulation)at a single dose.
Bioavailability | 5 days
  Relative bioavailability (secondarily measured by tmax and t1/2) between metformin hydrochloride 500 mg extended release caplet (test formulation) and metformin hydrochloride 500 mg prolonged release tablet (reference formulation)at multiple doses.
Adverse events | 2 months
  Adverse events occurred during the study conduct (2 months) were properly and sufficiently handled and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Danang A. Yunaidi, MD, Principal Investigator — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Caille G, Lacasse Y, Raymond M, Landriault H, Perrotta M, Picirilli G, Thiffault J, Spenard J. Bioavailability of metformin in tablet form using a new high pressure liquid chromatography assay method. Biopharm Drug Dispos. 1993 Apr;14(3):257-63. doi: 10.1002/bdd.2510140308. PMID 8490112
- [Background] Cheng CL, Chou CH. Determination of metformin in human plasma by high-performance liquid chromatography with spectrophotometric detection. J Chromatogr B Biomed Sci Appl. 2001 Oct 5;762(1):51-8. doi: 10.1016/s0378-4347(01)00342-5. PMID 11589458
- [Background] Najib N, Idkaidek N, Beshtawi M, Bader M, Admour I, Alam SM, Zaman Q, Dham R. Bioequivalence evaluation of two brands of metformin 500 mg tablets (Dialon & Glucophage)--in healthy human volunteers. Biopharm Drug Dispos. 2002 Oct;23(7):301-6. doi: 10.1002/bdd.326. PMID 12355581
- [Background] Scheen AJ. Clinical pharmacokinetics of metformin. Clin Pharmacokinet. 1996 May;30(5):359-71. doi: 10.2165/00003088-199630050-00003. PMID 8743335